CLINICAL TRIAL: NCT05267340
Title: Neural Mechanisms of Meditation Training in Healthy and Depressed Adolescents: An MRI Connectome Study PART 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 19-29083 (c); R33AT009864 (NIH)
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Depression Mild; Depression Moderate; Depression, Teen
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: TARA Training (Experimental): Behavioral: Training for Awareness, Resilience, and Action (TARA)
  This will be a 12-week group meditation training - Training for Awareness, Resilience, and Action (TARA)
  Interventions: Behavioral: TARA
- Control: Psycho-Education (Active Comparator): Behavioral: Training for Awareness, Resilience, and Action (TARA) without the mindfulness meditation components
  This will be a 12-week group meditation training - Training for Awareness, Resilience, and Action (TARA) without the mindfulness meditation components
  Interventions: Behavioral: Psycho-Education

INTERVENTIONS:
Behavioral: TARA — This will be a 12-week group meditation training - Training for Awareness, Resilience, and Action (TARA)
  Arms: Experimental: TARA Training
Behavioral: Psycho-Education — This will be a 12-week group meditation training - Training for Awareness, Resilience, and Action (TARA) without the mindfulness meditation components
  Arms: Control: Psycho-Education

SUMMARY:
The primary objective will be to study changes in putamen connectivity and depression severity in depressed teens with meditation training. H1: Putamen node strength will increase in the training group compared to the active controls. H2: This increase in node strength will correlate with practice amount recorded by participants. H3: There will be a significant reduction in self-rated depression symptoms following the training as measured by the Reynolds Adolescent Depression Scale (RADS-2), compared to controls. H4: This reduction will correlate with the increase in putamen node strength.

Design and Outcomes: The current research study design will utilize an individually randomized group treatment, open-label, active-controlled clinical trial to test the efficacy and safety of the investigator's innovative mindfulness meditation intervention (Training for Awareness Resilience and Action [TARA]) on the primary outcome (Putamen structural node strength) and secondary outcome (depression symptoms measured using Reynolds Adolescent Depression Scale [RADS-2]) in depressed adolescents between the ages of 14 to 18 years old.

ELIGIBILITY:
INCLUSION CRITERIA:

Female and male adolescents with elevated depression (RADS-2 T-score >50 or as judged by the study physician), 14-18 years old.

We will use Medical History form a (NCCIH Version 1.0). The required current status of participants within 4 weeks prior to randomization is absence of current medical, neurological, or psychiatric conditions except for a diagnosis of a DSM-5 depressive disorder (which is allowed but not required). Due to the exceptionally high comorbidity with depression and anxiety, participants with a depressive disorder and comorbid anxiety disorder will also be allowed to enter the study.

Fluency in English. Being under the care of a primary care provider or a mental health provider. Access to a smartphone, a tablet or a computer, on which program "Zoom" can be run for remote participation in the intervention.

EXCLUSION CRITERIA:

Subjects younger or older than 14-18 years old. Subjects who have a significant medical disorder or mental health disorder other than a DSM-5 depressive disorder or a depressive disorder with a comorbid anxiety disorder. We will use Phone Pre-Screener and Medical History form a (NCCIH Version 1.0) to exclude any adolescent who has been clinically diagnosed with any significant medical disorder that would prevent him or her from performing yoga-based movements (e.g., cerebral palsy), neurological disorder (e.g., multiple sclerosis, severe head trauma) or mental health disorder other than a DSM-5 depressive disorder or a DSM-5 depressive disorder and comorbid anxiety disorder (e.g., psychosis, schizophrenia, schizoaffective disorder, bipolar disorder, ADHD, autism spectrum disorder, anorexia nervosa, PTSD) or has intellectual disability, or suicidal ideation or attempt in past 3 months. (Please note that a diagnosis of a DSM-5 depressive disorder is allowed, but not required, to enter our study).

Subjects who are taking any psychotropic medication other than one of the first-line selective serotonin reuptake inhibitor (SSRI) antidepressant medications (i.e., fluoxetine, escitalopram, sertraline).

MRI contraindications (metallic objects on or inside the body, e.g., braces), some types of tatoos, and pregnancy.

Pregnancy or any plans to become pregnant during the study is an exclusion criterion for entrance into the study. Women of reproductive capability will be asked to employ at least one of the following allowable contraception methods until they complete their second MRI scan: birth control implant, birth control shot, birth control patch, birth control pill, condom, internal condom, birth control sponge, cervical cap, spermicide, fertility awareness (calendar method), outercourse and abstinence.

The study's pregnancy-related policy and procedure are as follows. First, all female participants will be asked to fill out a pregnancy screening questionnaire and then take a urine pregnancy test immediately prior to entering the MRI scanner room. Any subject that is either pregnant or might possibly be pregnant are not allowed to enter the MRI scanner room. Results of the urine pregnancy screening test will be shared with the adolescent subject only and not with the adolescent's parents or legal guardians. As per California state confidentiality laws, the results of pregnancy tests in minors cannot be shared with the minor's parent or legal guardian without the written permission of the minor. If the pregnancy test is positive, we will counsel the teen and give her referrals to teen pregnancy resources such as Planned Parenthood. If the participant is pregnant, the participant is not allowed to enter the study until the pregnancy is over. Second, if the participant who is in the intervention group becomes pregnant during the course of the study after the first MRI scan, she will be allowed to finish participating in the group intervention since there are no known potential adverse effects on the fetus due to meditation. However, although there are no known adverse negative effects of MRI scans on the fetus, we have decided to be conservative in our study and not allow participants who become pregnant during the study after the first MRI scan to have the second MRI scan in order to minimize any potential risk to the unborn fetus.

Not allowable: Current mindfulness training (e.g. MBSR, MBCT, DBT) and/or practice with a typically sitting meditation or yoga of 20 or more minutes two or more times per week within 60 days prior to study entry.

Potential adolescent subjects with current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to the study requirements will be excluded and not allowed to enter the study. We will use the Brief Screener for Tobacco, Alcohol, and other Drugs (BSTAD) developed by National Institute on Drug Abuse (NIDA) to determine higher risk subjects who will be excluded: https://www.drugabuse.gov/adolescent-substance-use-screening-tools.

Potential subjects with an inability or unwillingness to give written informed assent or whose legal guardian/representative are unable or unwilling to give written informed consent will be excluded and not allowed to enter the study.

Any other factors preventing from participation according to the judgment of the Principal Investigators.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change in Putamen node strength | Baseline/randomization and 12 weeks after baseline/randomization
  Change in the Putamen node strength assessed using diffusion MRI

SECONDARY OUTCOMES:
Change in Depression Symptoms | Baseline/randomization and 12 weeks after baseline/randomization
  Change in the score on the Reynold's Adolescent Depression Scale-2 (RADS-2). The RADS-2 has a possible range of 30 to 120. Higher scores represent higher levels of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Tony T Yang, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No